CLINICAL TRIAL: NCT03127696
Title: A Randomised Placebo-controlled Study of Fecal Microbiota Transplant (FMT) to Impact Body Weight and Glycemic Control in Obese Subjects With Type 2 Diabetes Mellitus
Brief Title: Randomised Placebo-controlled Study of FMT to Impact Body Weight and Glycemic Control in Obese Subjects With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMT-DM-RCT study
Record Dates: First submitted 2017-04-07; First posted 2017-04-25 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Type2 Diabetes; Type 2 Diabetes Mellitus; Obese
Keywords: Fecal Microbiota Transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Fecal Microbiota Transplantation; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FMT + LMP (Experimental): FMT and lifestyle modification program
  Interventions: Procedure: Fecal Microbiota Transplantation; Behavioral: Lifestyle Modification Program
- FMT alone (Experimental): Fecal Microbiota Transplantation
  Interventions: Procedure: Fecal Microbiota Transplantation
- Sham + LMP (Sham Comparator): Sham and lifestyle modification program
  Interventions: Behavioral: Lifestyle Modification Program; Procedure: Sham

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — FMT
  Arms: FMT + LMP; FMT alone
Behavioral: Lifestyle Modification Program — Lifestyle
  Arms: FMT + LMP; Sham + LMP
Procedure: Sham — Sham
  Arms: Sham + LMP

SUMMARY:
Faecal microbiota transplantation (FMT) represents a clinically feasible way to restore the gut microbial ecology, and has proven to be a breakthrough for the treatment of recurrent Clostridium difficile infection. Early results in human have shown that FMT from lean donor when transplanted into subjects with metabolic syndrome resulted in a significant improvement in insulin sensitivity and an increased in intestinal microbial diversity, including a distinct increase in butyrate-producing bacterial strains. The therapy is generally well tolerated and appeared safe. No clinical studies have assessed the efficacy of FMT in obese subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
There is a worldwide epidemic of obesity and type 2 diabetes mellitus. The prevalence of obesity and type 2 diabetes mellitus continues to rise at an alarming rate. Weight loss is associated with reductions in risk of morbidity and mortality from obesity. Conventional non-pharmacological interventions based on diet and exercise showed limited long-term success in producing sustained weight loss. Although obese patients with type 2 diabetes mellitus may be treated by medications or by bariatric surgery, these alternatives are limited by incomplete resolution of the diseases, high cost or potential surgical-related morbidity. Further research focusing on increasing effectiveness of interventions and new ways to achieve weight loss in these individuals are needed.

Recently, accumulating evidence supports a role of the enteric microbiota in the pathogenesis of obesity-related insulin resistance. Obesity is associated with changes in the composition of the intestinal microbiota, and the obese microbiome appears to be more efficient in harvesting energy from the diet. Colonization of germ-free mice with an 'obese microbiota' results in a significantly greater increase in total body fat than colonization with a 'lean microbiota', suggesting gut microbiota as an additional contributing factor to the pathophysiology of obesity. Obese and lean phenotypes can also be induced in germ-free mice by transfer of fecal microbiota from human donors. These data have led to the use of microbiota therapeutics as a potential treatment for metabolic syndrome and obesity.

Clinical trials are being conducted to evaluate its use for other conditions. Early results in human have shown that FMT from lean donor when transplanted into subjects with metabolic syndrome resulted in a significant improvement in insulin sensitivity and an increased in intestinal microbial diversity, including a distinct increase in butyrate-producing bacterial strains. The therapy is generally well tolerated and appeared safe. No clinical studies have assessed the efficacy of FMT in obese subjects with type 2 diabetes mellitus.

No clinical studies have assessed the efficacy of FMT in obese subjects with type 2 diabetes mellitus.

A subgroup of 30 subjects will be analyzed at week 24. The difference and proportion in microbiome in different arms, microbial factors, and trans-kingdom correlation of microbial engraftment will be correlated with clinical data in an unblinded manner.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70; and
* BMI >=28 kg/m2 and < 45 kg/m2; and
* A diagnosis of Type 2 diabetes mellitus for >=3 months; and
* Written informed consent obtained

Exclusion Criteria:

* Current pregnancy
* Use of any weight loss medications in the preceding 1 year
* Known history or concomitant significant gastrointestinal disorders (including Inflammatory Bowel Disease, current colorectal cancer, current GI infection)
* Known history or concomitant significant food allergies
* Immunosuppressed subjects
* Known history of severe organ failure (including decompensated cirrhosis), inflammatory bowel disease, kidney failure, epilepsy, acquired immunodeficiency syndrome
* Current active sepsis
* Active malignant disease in recent 2 years
* Known contraindications to oesophago-gastro-duodenoscopy (OGD)
* Use of probiotic or antibiotics in recent 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with at least 20% lean-associated microbiota in recipients after FMT compared with subjects receiving lifestyle intervention alone up to week 24 | 24 weeks
  Proportion of subjects with at least 20% lean-associated microbiota in recipients after FMT compared with subjects receiving lifestyle intervention alone up to week 24.

SECONDARY OUTCOMES:
Changes in microbial composition (including bacteriome and virome), function and metabolite | 4, 16, 20, 24 week
  Changes in microbial composition (including bacteriome and virome), function and metabolite at weeks 4, 16, 20 and 24 compared with baseline
Changes in microbiome of stool (including bacteriome and virome) | 4, 16, 24 week
  Changes in microbiome of stool (including bacteriome and virome) at weeks 4, 16 and 24 compared with baseline
Difference in microbiome (including bacteriome and virome) compared between subjects in different treatment arm | 24 week and 52 week
  Compare the difference in microbiome among different treatment arms
Proportion of microbiome (including bacteriome and virome) derived from recipient, donor or both in subjects who received FMT | weeks 4, 8, 12, 16, 20, 24 and 52
  Proportion of microbiome (including bacteriome and virome) derived from recipient, donor or both in subjects who received FMT
Difference in microbiome (including bacteriome and virome) compared between subjects who have weight loss and those do not have weight loss | weeks 4, 8, 12, 16, 20, 24 and 52
  Difference in microbiome (including bacteriome and virome) compared between subjects who have weight loss and those do not have weight loss
Microbial factors (including bacteriome and virome) that are associated with percentage of body weight loss | weeks 4, 8, 12, 16, 20, 24 and 52
  Microbial factors (including bacteriome and virome) that are associated with percentage of body weight loss
Trans-kingdom correlation of microbial engraftment | weeks 4, 8, 12, 16, 20, 24 and 52
  Trans-kingdom correlation of microbial engraftment after FMT between bacteriome, and virome
Proportion of subjects with serious adverse events compared between treatment arm, especially those related to FMT | weeks 4, 8, 12, 16, 20, 24 and 52
  Proportion of subjects with serious adverse events compared between treatment arm, especially those related to FMT
Explore changes in fungome microbiota | weeks 4, 8, 12, 16, 20, 24 and 52
  Explore changes in fungome microbiota
Proportion of subjects achieving at least 10% reduction in weight compared with baseline | 52 weeks
  Proportion of subjects achieving at least 10% reduction in weight at 52 weeks
Proportion of subjects achieving at least 10% reduction in weight compared with baseline | 24 weeks
  Proportion of subjects achieving at least 10% reduction in weight at 24 weeks
Changes in body weight to calculate body mass index (BMI) at weeks 24 and 52 compared with baseline | 24 week and 52 week
  Compare the change in weight to calculate the BMI among different treatment arms
Changes in biochemical parameters | 24 week and 52 week
  Changes in liver biochemistry, fasting glucose, fasting lipids, fasting insulin, HbA1C at weeks 24 and 52 compared with baseline
A 30% decrease in insulin resistance at weeks 24 compared with baseline | week 24
  A 30% decrease in insulin resistance at weeks 24 compared with baseline
Changes in liver stiffness to assess improvement of other metabolic disease weeks 24 compared with baseline | week 24
  Changes in liver stiffness to assess improvement of other metabolic disease weeks 24 compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Siew NG, Prof., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma RC, Lin X, Jia W. Causes of type 2 diabetes in China. Lancet Diabetes Endocrinol. 2014 Dec;2(12):980-91. doi: 10.1016/S2213-8587(14)70145-7. Epub 2014 Sep 10. PMID 25218727
- [Background] Haslam DW, James WP. Obesity. Lancet. 2005 Oct 1;366(9492):1197-209. doi: 10.1016/S0140-6736(05)67483-1. PMID 16198769
- [Background] Poobalan AS, Aucott LS, Smith WC, Avenell A, Jung R, Broom J. Long-term weight loss effects on all cause mortality in overweight/obese populations. Obes Rev. 2007 Nov;8(6):503-13. doi: 10.1111/j.1467-789X.2007.00393.x. PMID 17949355
- [Background] Dombrowski SU, Knittle K, Avenell A, Araujo-Soares V, Sniehotta FF. Long term maintenance of weight loss with non-surgical interventions in obese adults: systematic review and meta-analyses of randomised controlled trials. BMJ. 2014 May 14;348:g2646. doi: 10.1136/bmj.g2646. PMID 25134100
- [Background] Turnbaugh PJ, Hamady M, Yatsunenko T, Cantarel BL, Duncan A, Ley RE, Sogin ML, Jones WJ, Roe BA, Affourtit JP, Egholm M, Henrissat B, Heath AC, Knight R, Gordon JI. A core gut microbiome in obese and lean twins. Nature. 2009 Jan 22;457(7228):480-4. doi: 10.1038/nature07540. Epub 2008 Nov 30. PMID 19043404
- [Background] Turnbaugh PJ, Ley RE, Mahowald MA, Magrini V, Mardis ER, Gordon JI. An obesity-associated gut microbiome with increased capacity for energy harvest. Nature. 2006 Dec 21;444(7122):1027-31. doi: 10.1038/nature05414. PMID 17183312
- [Background] Ridaura VK, Faith JJ, Rey FE, Cheng J, Duncan AE, Kau AL, Griffin NW, Lombard V, Henrissat B, Bain JR, Muehlbauer MJ, Ilkayeva O, Semenkovich CF, Funai K, Hayashi DK, Lyle BJ, Martini MC, Ursell LK, Clemente JC, Van Treuren W, Walters WA, Knight R, Newgard CB, Heath AC, Gordon JI. Gut microbiota from twins discordant for obesity modulate metabolism in mice. Science. 2013 Sep 6;341(6150):1241214. doi: 10.1126/science.1241214. PMID 24009397
- [Background] Smith MI, Yatsunenko T, Manary MJ, Trehan I, Mkakosya R, Cheng J, Kau AL, Rich SS, Concannon P, Mychaleckyj JC, Liu J, Houpt E, Li JV, Holmes E, Nicholson J, Knights D, Ursell LK, Knight R, Gordon JI. Gut microbiomes of Malawian twin pairs discordant for kwashiorkor. Science. 2013 Feb 1;339(6119):548-54. doi: 10.1126/science.1229000. Epub 2013 Jan 30. PMID 23363771
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665
- [Background] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514
- [Background] Kelly CR, Kahn S, Kashyap P, Laine L, Rubin D, Atreja A, Moore T, Wu G. Update on Fecal Microbiota Transplantation 2015: Indications, Methodologies, Mechanisms, and Outlook. Gastroenterology. 2015 Jul;149(1):223-37. doi: 10.1053/j.gastro.2015.05.008. Epub 2015 May 15. PMID 25982290
- [Background] Kassam Z, Lee CH, Yuan Y, Hunt RH. Fecal microbiota transplantation for Clostridium difficile infection: systematic review and meta-analysis. Am J Gastroenterol. 2013 Apr;108(4):500-8. doi: 10.1038/ajg.2013.59. Epub 2013 Mar 19. PMID 23511459
- [Background] Wong SK, Kong AP, Mui WL, So WY, Tsung BY, Yau PY, Chow FC, Ng EK. Laparoscopic bariatric surgery: a five-year review. Hong Kong Med J. 2009 Apr;15(2):100-9. PMID 19342735
- [Background] Chan JC, So W, Ma RC, Tong PC, Wong R, Yang X. The Complexity of Vascular and Non-Vascular Complications of Diabetes: The Hong Kong Diabetes Registry. Curr Cardiovasc Risk Rep. 2011 Jun;5(3):230-239. doi: 10.1007/s12170-011-0172-6. Epub 2011 Apr 12. PMID 21654912
- [Background] Wong VW, Chan RS, Wong GL, Cheung BH, Chu WC, Yeung DK, Chim AM, Lai JW, Li LS, Sea MM, Chan FK, Sung JJ, Woo J, Chan HL. Community-based lifestyle modification programme for non-alcoholic fatty liver disease: a randomized controlled trial. J Hepatol. 2013 Sep;59(3):536-42. doi: 10.1016/j.jhep.2013.04.013. Epub 2013 Apr 23. PMID 23623998
- [Background] Wang S, Xu M, Wang W, Cao X, Piao M, Khan S, Yan F, Cao H, Wang B. Systematic Review: Adverse Events of Fecal Microbiota Transplantation. PLoS One. 2016 Aug 16;11(8):e0161174. doi: 10.1371/journal.pone.0161174. eCollection 2016. PMID 27529553
- [Derived] Ng SC, Xu Z, Mak JWY, Yang K, Liu Q, Zuo T, Tang W, Lau L, Lui RN, Wong SH, Tse YK, Li AYL, Cheung K, Ching JYL, Wong VWS, Kong APS, Ma RCW, Chow EYK, Wong SKH, Ho ICH, Chan PKS, Chan FKL. Microbiota engraftment after faecal microbiota transplantation in obese subjects with type 2 diabetes: a 24-week, double-blind, randomised controlled trial. Gut. 2022 Apr;71(4):716-723. doi: 10.1136/gutjnl-2020-323617. Epub 2021 Mar 30. PMID 33785557